CLINICAL TRIAL: NCT03546894
Title: An Observational Parallel Group Phase 4 Study to Determine Progression-Free Survival and Evaluate Patient Experience for Patients With Metastatic ALK+ Non-Small Cell Lung Cancer (NSCLC) Treated With ALK Inhibitors
Brief Title: A Study to Determine Progression-free Survival (PFS) and Evaluate Participant Experience for Participants With Metastatic Anaplastic Lymphoma Kinase-positive (ALK+) Non-Small Cell Lung Cancer (NSCLC) Treated With Anaplastic Lymphoma Kinase (ALK) Inhibitors
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: NSCLC-4001; U1111-1213-1757 (Registry Identifier: WHO)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Anaplastic Lymphoma Kinase-positive; Carcinoma Non-small-cell Lung
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib; alectinib; ceritinib; lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Brigatinib: The dosage and regimen of brigatinib (ALK inhibitors) will be decided by participant's prescribing physician and will not be determined by participation in the study.
  Interventions: Drug: Brigatinib
- Any FDA Approved ALK Inhibitor Other Than Crizotinib: The dosage, regimen of any Food and Drug Administration (FDA) approved ALK inhibitor (at any point in therapy) other than crizotinib will be decided by participant's prescribing physician and will not be determined by participation in the study.
  Interventions: Drug: Alectinib; Drug: Ceritinib; Drug: Lorlatinib; Drug: Any FDA Approved ALK Inhibitors

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablets.
  Groups: Brigatinib
Drug: Alectinib — Alectinib capsules.
  Groups: Any FDA Approved ALK Inhibitor Other Than Crizotinib
Drug: Ceritinib — Ceritinib capsules.
  Groups: Any FDA Approved ALK Inhibitor Other Than Crizotinib
Drug: Lorlatinib — Lorlatinib capsules.
  Groups: Any FDA Approved ALK Inhibitor Other Than Crizotinib
Drug: Any FDA Approved ALK Inhibitors — FDA approved ALK inhibitors available for treatment.
  Groups: Any FDA Approved ALK Inhibitor Other Than Crizotinib

SUMMARY:
The primary purpose of this study is to determine the differences in PFS for participants who have been receiving brigatinib as ALK inhibitor therapy for ALK+NSCLC compared to those participants receiving alectinib, ceritinib, lorlatinib, or other ALK inhibitors that may become available during study treatment.

DETAILED DESCRIPTION:
This is a prospective and non-interventional study of participants with ALK+NSCLC. The study will seek to determine the real-world differences in the PFS of participants taking brigatinib or any FDA approved ALK inhibitor other than crizotinib in routine clinical practice and will evaluate participant's quality of life, daily function, general condition, and treatment satisfaction.

The study will enroll approximately 160 participants: 80 participants taking brigatinib, and 80 participants taking FDA approved ALK inhibitors other than crizotinib. Participants will be enrolled in one of the 2 cohorts:

* Brigatinib
* Any FDA Approved ALK Inhibitor Other Than Crizotinib

This trial will be conducted in the United States. Upon enrollment into the study, participants will complete a study-specific baseline questionnaire and four validated instrument questionnaires. After that, participants will complete a study-specific monthly questionnaire and four validated instrument questionnaires, which will be made available to participants every 30 days. Participants will be sent automatic e-mail reminders every 30 days when new surveys become available. All participants will receive a notice on completion of their participation in the study at approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has ALK+ NSCLC.
2. Has been prescribed:

   * Brigatinib at any point in therapy, OR
   * Any FDA approved ALK inhibitor at any point in therapy other than crizotinib. Participants who were previously on crizotinib, but are now on another ALK inhibitor are eligible for study participation.
3. Has internet access.
4. Is willing to answer regular e-surveys and allow for the prescriber or clinic to provide data on the status of the participant's NSCLC.

Exclusion Criteria:

1. Has received any investigational compound within 90 days prior to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with ALK+NSCLC and who currently prescribed an ALK inhibitor, except crizotinib.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Prescriber-confirmed PFS | Baseline up to disease progression or death due to any cause, whichever comes first (approximately 24 months)
  PFS is defined as the time from the date of the first administration of ALK inhibitor to the date of the first documentation of disease progression or death due to any cause, whichever comes first. PFS will be based on prescriber confirmed progression. Participants that withdraw, drop out, or are lost to follow-up before documentation of the events will be censored at the last date at which the participant was determined to be progression-free.

SECONDARY OUTCOMES:
Quality of Life Status Using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire -Lung Cancer (EORTC QLQ-LC13) | Baseline up to treatment cessation or up to approximately 24 months
  EORTC QLQ-LC13 contains 13 questions to assess for: dyspnea, and a series of single items including pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Score of each item will range from 0 to 100, where 0 indicates no symptoms and 100 indicates worst possible symptoms.
Daily Function Status by M.D. Anderson Symptom Inventory - Lung Cancer (MDASI-LC) | Baseline up to treatment cessation or up to approximately 24 months
  The MDASI-LC Module includes 22 questions to assess the severity of multiple lung cancer-related symptoms and the impact of these symptoms on daily functioning. Symptom assessments include: pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, numbness/tingling, coughing, constipation, sore throat, general activity, mood, work, relations with others, walking, and enjoyment of life. Scores for each item range from 0 to 10, where 0 indicates no symptoms and 10 indicates worst possible symptoms.
General Condition Status Using EuroQol Research Foundation EQ-5D-5L | Baseline up to treatment cessation or up to approximately 24 months
  The EQ-5D-5L is a standardized non-disease-specific instrument for use as a measure of generic health status. It has 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Treatment Satisfaction Using the Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Baseline up to treatment cessation or up to approximately 24 months
  The TSQM-9 contains 9 items assessing the following 3 domains: effectiveness (3 items), convenience (3 items) and global satisfaction (3 items).
Participant-reported PFS | Baseline up to disease progression or death due to any cause, whichever comes first (approximately 24 months)
  PFS is defined as the time from the date of the first administration of ALK inhibitor to the date of the first documentation of disease progression or death due to any cause, whichever occurs first. PFS will be based on participant reported progression. Participants that withdraw, drop out, or are lost to follow-up before documentation of the events will be censored at the last date at which the participant was determined to be progression-free.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- EmpiraMed, Inc., Maynard, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60294db2bf003ab499b0??page=1&idFilter=NSCLC-4001